CLINICAL TRIAL: NCT06655584
Title: ENDOREV: A Solution to Reduce Anxiety During Gynecological Consultations in Patients With Suspected Endometriosis?
Acronym: ENDOREV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poissy-Saint Germain Hospital (Other)
Collaborators: French Interregional Group of Clinical Research and Innovation (Other)
Responsible Party: Principal Investigator, Elise LUNELLI, research nurse, Poissy-Saint Germain Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01166-41
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Suspected Endometriosis
Keywords: endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, controlled, open-label interventional study on two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Experimental Group A: The patient will be installed in a reception room and will benefit from Bliss DTx digital therapy via a video headset and an audio headset for a duration of 13 minutes
  Interventions: Device: Virtual reality headset Bliss DTX
- group B (No Intervention): Group B control: The patient will be installed in a reception room and will be seated and wait for the doctor to arrive (no material)

INTERVENTIONS:
Device: Virtual reality headset Bliss DTX — The patient will be installed in a reception room and will benefit from Bliss DTx digital therapy via a video headset and an audio headset for a duration of 13 minutes
  Arms: Group A

SUMMARY:
The aim of the research is to evaluate the effectiveness of virtual reality on the anxiety of patients with suspected endometriosis in gynecological consultation.

Indeed, several studies prove that patients in this situation are anxious. We would like to offer help in reducing anxiety in this case by means of digital therapy.

As part of this study, the equipment used will be "Bliss DTX". This is a non-drug digital therapy (digital therapeutics) already used in various hospital departments.

Bliss DTX immerses patients in sound and image programs scientifically developed for their effect on pain and anxiety, mobilizing their abilities and placing them in an altered state of consciousness. Bliss DTX software is delivered to patients via a dedicated video headset (virtual reality) and audio headset, as part of an integrated solution.

Conduct of the study:

The patient will be taken care of on the day of the consultation by a clinical research nurse. It will be installed in a reception room in the consultation room. The nurse will give him a questionnaire on anxiety to complete before the consultation.

A draw will be carried out with two options:

1. Bliss DTX digital therapy via audio and video headphones lasting 13 minutes
2. Installation in the reception room while waiting for the doctor to arrive. After the consultation, the patient will complete a new questionnaire on her state of anxiety and her feelings during the consultation.

A telephone call will be made 6 months after the consultation to collect post-consultation information.

Duration :

Duration of 6 months on 46 patients followed for 18 months. Expected benefits

* Reduction of anxiety after consultation by diversion of attention
* Strengthening the bond of trust between the patient and the care team
* Better monitoring and better compliance with treatment and medical examinations
* Better pain management
* Improved quality of life

Possible side effects:

No particular risks or constraints, however, a virtual reality headset can cause symptoms such as: nausea, dizziness, sweating, paleness, balance disorders grouped under the term "cybernetosis" as well as epileptic seizures in people. subjects predisposed to convulsions.

DETAILED DESCRIPTION:
Title :

ENDOREV: A solution to reduce anxiety during gynecological consultations in patients with suspected endometriosis?

Description of the study :

Single-center, randomized, controlled, open-label interventional study on two parallel groups Study composed of 46 patients randomized into two groups A and B with a ratio of 1:1 Experimental Group A: The patient will be installed in a reception room and will benefit from Bliss DTx digital therapy via a video headset and an audio headset for a duration of 13 minutes Group B control: The patient will be seated and wait for the doctor to arrive (no material) The duration of inclusion is 18 months and individual participation is 6 months, that is to say 24 months for the entire study.

Completion of the questionnaire (IASTA Y-1) for both groups before the consultation and data collection.

Filling of the CRF in consultation by the doctor Completion of the questionnaire (IASTA Y-1) for both arms after the consultation and data collection Telephone call at 6 months with data collection on compliance with endometriosis monitoring

Objectives :

Primary objectives :

• Evaluate the effectiveness of virtual reality on anxiety in women with suspected endometriosis during the gynecological consultation.

Secondary objectives :

* Study the effect of virtual reality on compliance with endometriosis monitoring following the gynecological consultation
* Evaluate the effect of virtual reality on the pain felt during the gynecological examination
* Evaluate the level of satisfaction with the device during the session

Hypothesis :

* Null hypothesis (H0): No significant difference between groups on post-consultation anxiety scores after adjustment for pre-consultation anxiety scores
* Alternative hypothesis (H1): There is a significant difference between groups on post-consultation anxiety scores after adjustment for pre-consultation anxiety scores.

Inclusion criteria :

* Patient between 18 and 45 years old
* Patient referred for suspected endometriosis
* Patient consulting for the first time in the hospital
* Patient with first-line or second-line imaging documenting endometriosis (ultrasound or MRI)
* Patient agreeing to participate in the study and having signed informed consent
* Patient affiliated to a social security scheme
* Patient able to read and write French

Exclusion criteria:

* Patient with a history of major pelvic surgery for endometriosis
* Patient undergoing hysterectomy
* Virgin patient
* Pregnant woman
* Patient with psychiatric pathology
* Patient suffering from proven epilepsy
* Patient under judicial protection
* Patient under guardianship or curatorship
* Patient with visual or hearing impairment
* Patient with a progressive pathology responsible for chronic pain

Place of the study :

Intercommunal Hospital Center of Poissy Saint-Germain-En-Laye

Contact details :

Intercommunal Hospital Center of Poissy Saint-Germain-En-Laye Address: 10 rue du Champ Gaillard, 78300 Poissy Tel: +33139274581 Email: elise.lunelli@ght-yvelinesnord.fr

Speakers :

* Promoter: Intercommunal Hospital Center of Poissy Saint-Germain-En-Laye
* Coordinating investigator: Ms. Elise LUNELLI (registered nurse)

Funding :

GIRCI IDF and ARS IDF funding as part of the call for projects " Appel à projets recherche en soins (APRESO) "2024

Calendar :

Primary submission : 11/09/24 Secondary submission :26/09/24

ELIGIBILITY:
Inclusion Criteria:

* • Patient between 18 and 45 years old

  * Patient referred for suspected endometriosis
  * Patient consulting for the first time in the hospital
  * Patient with first-line or second-line imaging documenting endometriosis (ultrasound or MRI)
  * Patient agreeing to participate in the study and having signed informed consent
  * Patient affiliated to a social security scheme
  * Patient able to read and write French

Exclusion Criteria:

* • Patient with a history of major pelvic surgery for endometriosis

  * Patient undergoing hysterectomy
  * Virgin patient
  * Pregnant woman
  * Patient with psychiatric pathology
  * Patient suffering from proven epilepsy
  * Patient under judicial protection
  * Patient under guardianship or curatorship
  * Patient with visual or hearing impairment
  * Patient with a progressive pathology responsible for chronic pain

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants showing a reduction in post-consultation anxiety | Pre-consultation until post-consultation

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud FAUCONNIER, PROFESSOR, Study Chair — Pr FAUCONNIER
Locations (1):
- Poissy-Saint Germain Hospital, Poissy, France

IPD SHARING:
Plan to Share IPD: No
In accordance with the provisions of the law relating to data processing, files and freedoms (law 78-17 of January 6, 1978 as amended) and the general data protection regulation (EU) 2016/679 (GDPR), the patient has a right to object at any time to the processing of their data.